CLINICAL TRIAL: NCT00695695
Title: The Role of Hope in Adaptation to Uncertainty: The Experience of Caregivers of Children With Down Syndrome
Brief Title: The Experience of Caregivers of Children With Down Syndrome
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908142; 08-HG-N142
Record Dates: First submitted 2008-06-11; First posted 2008-06-12 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-02-03

CONDITIONS: Down Syndrome
Keywords: Parents; Down Syndrome; Hope; Uncertainty; Adaptation; DS; Survey
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will explore how caregivers adjust to having a child with Down syndrome.

Primary caregivers 18 years of age and older of a child with Down syndrome may be eligible for this study. Participants complete a 20- to 30-minute survey that explores the subject s thoughts and feelings about being a caregiver to a child with Down syndrome. Questions explore the impact on the subject of being a caregiver for a child with Down syndrome, the subject s uncertainties related to the child s condition and goals for the child related to social skills, behavior, learning and education, physical and mental health, independence, and other goals. It also asks questions about the caregiver, the family and the child with Down syndrome.

...

DETAILED DESCRIPTION:
The proposed study aims to explore the relationships between perceived uncertainty, hope and adaptation in caregivers of children with Down Syndrome (DS). There are often uncertainties surrounding the prognosis of DS which extend into various aspects of the child s life. In addition to the possibility of chronic medical conditions associated with the syndrome, there is also uncertainty related to the level of independence and cognitive, social and behavioral functioning that the child will achieve. It is not fully understood how caregivers adapt to having a child with DS in light of the uncertainty and the particular challenges associated with this condition. While a high level of perceived uncertainty may be seen as a threat to adaptation, there is also evidence that caregivers may find benefits in uncertainty. Literature suggests that a person s level of hope influences how the perceived uncertainty is appraised and that hope is also related to the process of adaptation. There is no research that systematically explores the relationship between perceived uncertainty, hope, and adaptation. This study s conceptual framework is based on Lazarus & Folkman s Transactional Model of Stress and Coping and is also informed by Snyder s conceptualization of hope and Mishel s theory of perceived uncertainty in illness. A cross-sectional research design will quantitatively explore the relationships between perceived uncertainty, hope, and adaptation. In addition, an open-ended section will be included to qualitatively describe the focus of caregivers hope for their child and how the focus of hope relates to the degree of hope. Participants will be recruited from DS support groups, website postings, listservs, and clinic patient lists. They will have the option of completing either a paper or online version of the survey, or completing the survey by phone. The main outcome variable is psychological adaptation to being a care giver for a child with DS.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be men and women ages 18 or older who are the primary caregivers of a child with Down syndrome. The parent may be a biological or adoptive parent or other primary caregiver and the child must reside with the primary caregiver.

EXCLUSION CRITERIA:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2008-05-14; Study Completion 2014-02-03

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Davis B. Mediators of the relationship between hope and well-being in older adults. Clin Nurs Res. 2005 Aug;14(3):253-72. doi: 10.1177/1054773805275520. PMID 15995154
- [Background] Folkman S, Greer S. Promoting psychological well-being in the face of serious illness: when theory, research and practice inform each other. Psychooncology. 2000 Jan-Feb;9(1):11-9. doi: 10.1002/(sici)1099-1611(200001/02)9:13.0.co;2-z. PMID 10668055
- [Background] Lipinski SE, Lipinski MJ, Biesecker LG, Biesecker BB. Uncertainty and perceived personal control among parents of children with rare chromosome conditions: the role of genetic counseling. Am J Med Genet C Semin Med Genet. 2006 Nov 15;142C(4):232-40. doi: 10.1002/ajmg.c.30107. PMID 17068805